CLINICAL TRIAL: NCT02002299
Title: Prospective Study of Colorectal Cancer Comparing the Surface With the Invasive Front
Brief Title: Does Surface Tell us About the Invasive Front in Colorectal Cancer
Acronym: CRC1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CRCtopfront1
Record Dates: First submitted 2013-08-02; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; surface; invasive front; tumor budding
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples Without DNA — Surgical resection specimens of colorectal cancers
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the invasive front in growth mode (expanding or infiltrative) and dedifferentiation (tumor budding) and comparing these with the tumor surface (polypose or flat) + / - ulceration in surgical specimens at colorectal cancer.

DETAILED DESCRIPTION:
Timetable: From 1 August 2013 to 31 July 2014.

Organisational arrangements: The project is deleted from the pathology department, Roskilde Hospital, and surgical department, Roskilde Hospital.

inclusion criteria All colorectal surgical specimens having cancer were the patient did not receive neoadjuvant treatment received in the pathology department in accordance with current guidelines with the cutting of the tumor area in parallel slices and photographed, so there is macroscopic photo documentation.

Microscopic tumors classified as adenocarcinoma of glandular type, mucinous adenocarcinoma, signet ring cell carcinoma.

When the specimens is received at the department of pathology and is included in the study the pathologist report is registered in a local database.

ELIGIBILITY:
Inclusion Criteria:

* All surgical preparations from patients with colorectal cancer that did not receive neoadjuvant treatment received in the pathology department in accordance with current guidelines with the cutting of the tumor area in parallel slices and photographed, so there is macroscopic photo documentation.

Microscopic tumors classified as adenocarcinoma of glandular type, mucinous adenocarcinoma, signet ring cell carcinoma.

Exclusion Criteria:

* All surgical preparations from patients with colorectal cancer where the patient received neoadjuvant therapy or when surgery preparation could not be received by current guidelines and all preparations where it is not possible to obtain macroscopic image of the parallel slices.

Microscopic tumors that can not be classified as adenocarcinoma of the glandular type, mucinous adenocarcinoma or signet ring cell carcinoma excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients from Roskilde Hopsital with colorectal cancer who is having surgical resection of the tumor
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
invasive front growth pattern | The histopathological study for one specimens takes one week at average, results will be published shortly after july 2014 (one year after start)
  Microscopic divided tumors after growth pattern at the invasive front (tumor-bottom), rated on average, there is immunohistochemical stained for pancytokeratin. A points 1-4 described by Franzen et al (2008) used: tumor bottom is regular and smooth (score 1), tumor-bottom is irregular with large cell clusters (score 2), tumor-bottom is irregular with large and small clusters (score 3) and tumor-bottom consists almost entirely of smaller clusters (score 4).
  It is also noted whether there is a tumor budding or not. Tumor budding is a histological phenomenon that reflect loss of adhesion between tumor cells in the stroma of the invasive front of colorectal cancers. It is present if more than five groups containing 1-4 cancer cells each, within a microscopic area on x20 (Uneo et al (x25), 2002 and Mitrovic et al (x20), 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Eiholm, MD, Principal Investigator — Department of Pathology, Roskilde Hospital, Denmark
Locations (1):
- Department of Pathology,, Roskilde, Roskilde, Denmark